CLINICAL TRIAL: NCT05421754
Title: Low Burden Wearable Sensor System for Diagnosing Obstructive Sleep Apnea Over Multiple Nights: Diagnostic Agreement With Home Sleep Testing
Brief Title: ANNE Diagnostic Agreement With Home Sleep Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Sibel Health Inc. (Industry)
Responsible Party: Principal Investigator, Phyllis Zee, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU00214445
Record Dates: First submitted 2022-06-09; First posted 2022-06-16 (Actual); Results first posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Intervention Model Description: Patients will use ANNE Sleep system with Home Sleep Testing (HST) during one night followed by three subsequent nights with the ANNE Sleep system alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ANNE Sleep (Experimental): After consent, subjects will wear the ANNE Sleep system with HST for 1 night and 3 nights with ANNE sleep system alone.
  Interventions: Device: ANNE Sleep

INTERVENTIONS:
Device: ANNE Sleep — ANNE Sleep system for 1 night with HST followed by 3 nights of ANNE Sleep system alone.

SUMMARY:
The main objective of this study is to provide an adequately powered study that would provide evidence on the non-inferiority of ANNE to a Home Sleep Test (HST).

DETAILED DESCRIPTION:
The main objective of this study is to provide an adequately powered study that would provide evidence on the non-inferiority of ANNE to a Home Sleep Test (HST) for the diagnosis of moderate to severe OSA.

Other study objectives include:

* Determining diagnostic yield from multiple nights and better usability compared to current HST in the intended population. This will include all subjects and a focus on olders 65 and older.
* Gathering participant feedback on the use of the sensors and use of the application elicited through focus groups

ELIGIBILITY:
Inclusion Criteria:

* 22 years old.

  * Subjects with suspected OSA based on history and physical. Subjects with self-reported symptoms of OSA based on the STOP-Bang questionnaire indicating affirmative answers to any of the following: snoring, daytime fatigue/sleepiness/tiredness, partners who have observed the subject stopping breathing or choking/gasping during sleep. Persons with a previous diagnosis of OSA are also eligible.
  * Willingness to give written consent and comply with study procedures

Exclusion Criteria:

-An unstable medical condition, acute or chronic, that in the opinion of the investigator puts the subject at health risks related to this trial or interferes with the clinical trial and data collection based on the opinion of the investigator, this includes but is not limited to: A. Significant cardiorespiratory disease: patients that are oxygen dependent, previous hospitalization for cardiorespiratory issues, or left ventricular ejection fraction ≤ to 40% B. Respiratory muscle weakness due to a neuromuscular condition C. Awake hypoventilation or suspicion of sleep related hypoventilation D. Chronic opioid medication use E. History of stroke F. History of severe insomnia

* Inability to understand instructions
* Has a skin abnormality that precludes assessment
* Has a history of dementia
* Patients with implanted pacemakers or defibrillators

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Data stored and used for future research will be de-identified. Data will not be used for future research outside of the scope of this study.

REFERENCES:
- [Derived] Walter J, Lee JY, Blake S, Kalluri L, Cziraky M, Stanek E, Miller J, Harty BJ, Yu L, Park J, Zhang M, Coughlin S, Serao A, Lee J, Buban A, Bae M, Edel C, Toloui O, Rangel SM, Power T, Xu S. A new wearable diagnostic home sleep testing platform: comparison with available systems and benefits of multinight assessments. J Clin Sleep Med. 2023 May 1;19(5):865-872. doi: 10.5664/jcsm.10432. PMID 36692166

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-eight participants consented to the study and thirty participants started the study. Eight participants decided not to participate before any study procedures or were lost to follow-up after the consent process.
Period: Overall Study
Arm/Group | ANNE Sleep
Started | 30
Completed | 29
Not Completed | 1
Not completed — Technical issue with sensor | 1

BASELINE CHARACTERISTICS:
Arm/Group | ANNE Sleep
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (15.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 10
  Sex: Male | 17
  Sex: Did not answer | 3
Race/Ethnicity, Customized [Number; unit: participants] — Participants could indicate more than one race.
  participants
    Race : Asian | 8
    Race : Black or African American | 1
    Race : White | 19
    Race : Did not answer | 3
    Race : Hispanic or Latino | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.2 (3.9)
Epworth Sleepiness Scale [Median (Inter-Quartile Range); unit: units on a scale] — Epworth Sleepiness Scale is a self-administered questionnaire to provide a measurement of the subject's general level of daytime sleepiness. Subject rate on a scale of 1-3 for each of the eight questions: 0= would never doze, 1=slight chance of dozing, 2=moderate change of dozing, and 3=high chance of dozing. The answers are added together to give a final score from 0 to 24, 24 being the highest level of daytime sleepiness. Scores of 16 or higher indicates a high level of daytime sleepiness.
  units on a scale | 8 [6 to 14]
Hypertension [Count of Participants; unit: Participants] | 8
Type II Diabetes [Count of Participants; unit: Participants] | 2
Asthma [Count of Participants; unit: Participants] | 2
Depression [Count of Participants; unit: Participants] | 6
Anxiety [Count of Participants; unit: Participants] | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent Agreement of ANNE Sleep System to Home Sleep Test (WatchPAT) for Diagnostic Performance to Detect Moderate to Severe Obstructive Sleep Apnea.
Description: To determine the percent agreement between the ANNE sleep system to a Home Sleep Test (WatchPAT) for diagnostic performance to positively detect moderate to severe obstructive sleep apnea.. The WatchPAT system and ANNE sleep were worn for a single night together. The ANNE sleep system was additionally analyzed for up to 3 multiple nights and the data from those nights was pooled to compare against WatchPAT system for positively detecting moderate to severe obstructive sleep apnea.
Time Frame: 4 nights
Measure: Number (95% Confidence Interval); unit: percent agreement
Arm/Group | ANNE Sleep
Number analyzed (Participants) | 29
percent agreement
  Single night | 58 [28 to 85]
  Multiple nights | 75 [42.8 to 94.5]

ADVERSE EVENTS:
Time Frame: Four nights
Arm/Group | ANNE Sleep
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT05421754/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT05421754/ICF_001.pdf